CLINICAL TRIAL: NCT03363893
Title: A Modular, Multipart, Multiarm, Open-label, Phase I/II Study to Evaluate the Safety and Tolerability of CT7001 Alone and in Combination With Anti-cancer Treatments in Patients With Advanced Malignancies
Brief Title: Modular Study to Evaluate CT7001 Alone in Cancer Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Carrick Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT7001_001; 2017-002026-20 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2017-12-06 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Malignancies
Keywords: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: Modular design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Module 1 Part A Multiple ascending dose cohort and Paired Biopsy Breast Cancer Expansion Cohort (Experimental): Module 1 Part A Multiple ascending dose cohort: Participants with advanced solid tumours receive CT7001 (samuraciclib) as oral monotherapy, in ascending dose cohorts, to identify the maximum tolerated dose (MTD), minimally biologically active dose (MBAD) and recommended dose for Phase II testing (RP2D).
  Following completion of the dose escalation part of Module 1A, participants to receive safe, tolerable and MBAD of CT7001 for the paired biopsy expansion cohort.
  Module 1 Part A Paired Biopsy Breast Cancer Expansion Cohort: Participants with locally advanced or metastatic breast cancer will receive CT7001 (samuraciclib) as oral monotherapy at the minimally biologically active dose (MBAD) and recommended dose for Phase II testing (RP2D).
  Interventions: Drug: CT7001
- Module 1 Part B-1 Triple-negative breast cancer (TNBC) Expansion (Experimental): Participants with locally advanced or metastatic triple-negative breast cancer (TNBC) will receive CT7001(samuraciclib) as oral monotherapy at the dose, frequency and schedule recommended from Module 1 Part A.
  Interventions: Drug: CT7001
- Module 1 Part B-2 Castrate resistant prostate Cancer (CRPC) Expansion (Experimental): Participants with castrate resistant prostate cancer will receive CT7001(samuraciclib) as oral monotherapy at the dose, frequency and schedule recommended from Module 1 Part A.
  Interventions: Drug: CT7001
- Module 2 Part A (Experimental): Participants with locally advanced or metastatic HR+ve and HER2-ve breast cancer will receive CT7001 (samuraciclib) at the dose, frequency and schedule recommended from Module 1 part A and will receive Fulvestrant solution in pre-filled syringe for intramuscular (IM) injection
  Interventions: Drug: CT7001; Drug: Fulvestrant
- Module 4 (Experimental): Participants with advanced solid tumours will receive CT7001(samuraciclib) oral monotherapy in a randomized, balanced, single-dose, two-treatment (fed v fasting), two-period, two-sequence crossover study followed by once daily continuous dosing.
  Interventions: Drug: CT7001

INTERVENTIONS:
Drug: CT7001 — Cyclin-dependent kinase 7 (CDK7) inhibitor given orally once daily until disease progression
  Other Names: Samuraciclib
Drug: Fulvestrant — Administered as 2 x 250mg intramuscular (IM) gluteal injections on Day 1, Day 15, Day 28 and every 28 days thereafter.
  Other Names: Faslodex
  Arms: Module 2 Part A

SUMMARY:
This is a modular, Phase I/II, multicentre study to investigate CT7001 monotherapy in advanced solid malignancies and to further investigate CT7001 as monotherapy or in combination with standard therapy in specific participant groups with Triple Negative Breast Cancer (TNBC), Castrate Resistant Prostate Cancer (CRPC) and in combination with fulvestrant for patients with hormone receptor-positive (HR+ve) / human epidermal growth factor-2 negative (HER2-ve) breast cancer.

DETAILED DESCRIPTION:
Module 1 comprises two sequential parts:

* Part A: First-in-human (FiH) dose escalation investigating the safety and tolerability of CT7001 to identify the minimum biologically active dose (MBAD) and maximum tolerated dose (MTD). Part A also includes a cohort expansion for breast cancer participants only: this includes sequential tumour biopsies for evaluation of pharmacokinetic (PK), pharmacodynamic (PD) and tumour responses. The module is completed.
* Part B: To refine the safety, tolerability, and PK and PD profiles of CT7001 monotherapy in participants with advanced solid malignancies from up to four tumour- specific cohorts, which may include, but is not limited to, triple-negative breast cancer, ovarian cancer, small-cell lung cancer and prostate cancer.

  * Part B, Cohort 1, Triple-Negative Breast Cancer (M1B-1 TNBC) treated with CT7001 as monotherapy. The module is completed.
  * Part B, Cohort 2, Prostate Cancer (M1B-2 CRPC) treated with CT7001 as monotherapy. The module is completed.
* Module 2 is a Phase Ib/II, 3-part safety and efficacy study in participants with hormone- receptor positive (HR+ve) and human epidermal growth factor-2 negative (HER2-ve) breast cancer. This module includes dosing CT7001 in combination with fulvestrant. Module 2 was planned to comprise of 3 parts; Part A (open-label, single-arm, ascending dose study), Part B (double blinded, randomised, placebo-controlled study) and Part C (crossover from Part B). However, only Module 2 Part A was initiated and completed. Therefore, further sections of this record only reflect Module 2 Part A information.
* Module 4 is a study investigating the effect of food on the PK of CT7001 monotherapy in participants with advanced solid malignancies. The module is completed.
* Module 6 was planned as a Phase 1 study to explore the tolerability of, and the total and peak exposure of, an enteric capsule formulation of CT7001 [CT7001(EC)], when given as monotherapy to patients with advanced solid malignancies. Module 6 was not initiated.

ELIGIBILITY:
Core Inclusion Criteria:

1. ECOG performance status 0 or 1 with no deterioration over the previous 2 weeks
2. Estimated life expectancy of greater than 12 weeks
3. Ability to swallow and retain oral medication
4. Women either of non-childbearing potential or of childbearing potential willing to practice effective contraception for the duration of the study and for 6 months (Module 1, Module 4) and 24 months (Module 2) after the last dose of CT7001
5. Sexually active male patients must be willing to use condoms with all sexual partners for the duration of the study and for 3 months after the last dose of CT7001.
6. Provision of signed and dated, written informed consent

Core Exclusion Criteria:

1. Any other malignancy that has been active or treated within the past 3 years, with the exception of cervical intraepithelial neoplasia and non-melanoma skin cancer
2. Any unresolved toxicity (except alopecia) from prior therapy of ≥ CTCAE Grade 2
3. Spinal cord compression or brain metastases, unless asymptomatic, stable, and not requiring steroids for at least 4 weeks before the first dose of investigational product (IP)
4. Refractory nausea and vomiting, chronic gastrointestinal (GI) disease or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of CT7001
5. Uncontrolled seizures
6. Active infection requiring systemic antibiotic, antifungal, or antiviral medication
7. Severe or uncontrolled medical condition or psychiatric condition
8. Active bleeding diatheses
9. Renal transplant
10. Known hepatitis B, hepatitis C, or human immunodeficiency virus infection
11. Breastfeeding or pregnancy
12. Receipt of systemic cytotoxic treatment for the malignancy within 28 days or ≤ 5 half-lives, whichever is shorter before the first dose of IP
13. Receipt of non-cytotoxic treatment for the malignancy within 5 half-lives of the drug before the first dose of IP
14. Receipt of corticosteroids (at a dose > 10 mg prednisone/day or equivalent) within 14 days before the first dose of IP
15. Receipt of any small-molecule investigational medicinal product (IMP) within 28 days or ≤ 5 half-lives, whichever is shorter before the first dose of IP
16. Receipt of any biological IMP (e.g., immune checkpoint blockers, antibodies, nanoparticles) within 42 days before the first dose of IP
17. Receipt of St John's Wort within 21 days before the first dose of IP or of another concomitant medication, herbal supplement, or food that is a strong inhibitor or inducer of CYP3A4, CYP2C19, CYP2D6, or P-glycoprotein (PGP) activity within 14 days before the first dose of CT7001
18. Receipt of a blood transfusion (blood or blood products) within 14 days before the first dose of IP
19. Known hypersensitivity to CT7001 or any excipient of the product
20. Impaired hepatic or renal function as demonstrated by any of the following laboratory values:

    1. Albumin < 30 g/L
    2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × the upper limit of normal (ULN)
    3. > 5.0 × ULN for patients with liver metastases
    4. Total bilirubin > 1.5 × ULN
    5. Serum creatinine > 1.5 × ULN
21. Liver function deteriorating in a manner that would likely make the participant meet the AST, ALT, or bilirubin levels specified above at the time of the first dose of IP
22. Other evidence of impaired hepatic synthesis function
23. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count (ANC) < 1.5 × 10^9/L
    2. Platelet count < 100 × 10^9/L
    3. Haemoglobin < 90 g/L
24. Persistent (> 4 weeks) severe pancytopenia due to previous therapy rather than to disease (ANC < 0.5 × 10^9/L or platelets < 50 x 10^9/L)
25. Cardiac dysfunction (defined as myocardial infarction within 6 months of study entry, New York Heart Association Class II/III/IV heart failure, unstable angina, unstable cardiac arrhythmias, or left ventricular ejection fraction < 55 percent)
26. Mean resting QT interval corrected for heart rate by the Fridericia formula (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs) obtained within 5 minutes of each other prior to the first dose
27. Any clinically important abnormalities in rhythm, conduction, or morphology on resting ECG (e.g., complete left bundle branch block, third degree heart block). Controlled atrial fibrillation (AF) is permitted
28. Any factor that increases the risk of QTc prolongation or of arrhythmic events (e.g., heart failure, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age)
29. In the opinion of the Investigator, unlikely to comply with study procedures, restrictions, or requirements
30. A history of haemolytic anaemia or marrow aplasia
31. Has received a live-virus vaccination within 28 days or less of planned treatment start

Additional Module 1A Inclusion Criteria:

1. Histological, radiological or cytological confirmation of an advanced non-haematological malignancy not considered to be appropriate for further standard treatment
2. Module 1A biopsy cohort only : at least one tumour suitable for repeat biopsy

Additional Module 1A Exclusion Criteria:

1. International normalised ratio (INR) ≥1.5

Additional Module 1B Inclusion Criteria

1. Histological or cytological confirmation of metastasis or locally advanced tumour
2. At least one line of systemic anti-cancer therapy
3. Disease measurable by RECIST v1.1

Additional Module 1B-1 (TNBC Expansion) Inclusion Criteria:

1. Histologically-confirmed carcinoma of breast not expressing oestrogen receptor (ER) or progesterone receptor (PR) and negative for human epidermal growth factor receptor 2 (HER2)
2. Documented disease progression on or within 6 months of most recent cytotoxic prior cytotoxic chemotherapy
3. Disease measurable by RECIST v1.1
4. Must have received at least one cytotoxic chemotherapy for metastatic/locally advanced disease

Additional Module 1B-1 (TNBC Expansion) Exclusion Criteria:

1. No more than three lines of cytotoxic chemotherapy for metastatic/locally advanced disease
2. No advanced, symptomatic visceral metastases
3. No known symptomatic central nervous system (CNS) metastases, carcinomatous meningitis or leptomeningeal disease
4. Prior exposure to CT7001
5. Patients who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are Carrick employees directly involved in the conduct of the trial

Additional Module 2A Inclusion Criteria:

1. Women only
2. Pre- or peri-menopausal women must have initiated LHRHa at least 28 days prior to first dose of CT7001/placebo
3. Histologically-confirmed, metastatic or locally advanced, ER+ve and/or PGR+ve and HER2-ve breast cancer
4. Disease measurable by RECIST v1.1
5. Documented objective disease progression while on, or within 6 months after the end of, the most recent therapy
6. Must have received an aromatase inhibitor together with a CDK4/6 inhibitor in the same line of therapy for locally advanced or metastatic disease or for treatment of early breast cancer if the disease-free interval was <12 months.
7. Ability to receive intramuscular injections.

Additional Module 2A Exclusion Criteria:

1. Prior therapy with fulvestrant
2. More than 2 lines of endocrine treatment for locally advanced or metastatic disease
3. Prior treatment with more than one line of cytotoxic chemotherapy for locally advanced or metastatic breast cancer.
4. Patients with liver metastasis will be limited to approximately 30-40% of the enrolled patients. l
5. Known hypersensitivity to CT7001, fulvestrant or any excipient of the investigational products
6. Patients who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are Carrick employees directly involved in the conduct of the trial

Additional Module 4 Inclusion Criteria:

1. Patients must be able to eat a high-fat meal, as provided by the study site, within a 30-minute period
2. Histological, radiological or cytological confirmation of an advanced non-haematological malignancy not considered to be appropriate for further standard treatment

Additional Module 4 Exclusion Criteria:

1. Patients who were unable to fast for at least 10 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events and Laboratory Abnormalities (Safety and Tolerability) | Screening to end of study
  Type, incidence and severity

SECONDARY OUTCOMES:
Maximum Plasma Concentration of CT7001 (and Fulvestrant, where applicable) (Cmax) | After the first dose and during the dosing period
  Cmax is the maximum observed plasma concentration of CT7001 (and Fulvestrant in Module 2 Part A) following oral dosing
Area Under the Curve (AUC) | After the first dose and during the dosing period
  Area under the plasma concentration-time curve representing the total drug exposure over time
Anti-tumour Activity according to RECIST v1.1 | Baseline until disease progression or withdrawal from the study
  Antitumour activity endpoints will be analysed using the evaluable for Response population based on RECIST assessment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, MBChB PhD, Principal Investigator — The Christie Hospital, Manchester, UK
Locations (23):
- United States (12):
  - Research Site 54, Tucson, Arizona
  - Research Site 31, Beverly Hills, California
  - Research Site 37, Tampa, Florida
  - Research Site 38, Chicago, Illinois
  - Research Site 34, Boston, Massachusetts
  - Research Site 47, Cincinnati, Ohio
  - Research Site 39, Columbus, Ohio
  - Research Site 36, Portland, Oregon
  - Research Site 44, Austin, Texas
  - Research Site 46, Dallas, Texas
  - Research Site 48, Salt Lake City, Utah
  - Research Site 33, Salem, Virginia
- United Kingdom (11):
  - Research site 11, Brighton
  - Research site 5, Cambridge
  - Research Site 7, Glasgow
  - Research Site 10, Liverpool
  - Research Site 9, London
  - Research Site 8, London
  - Research Site 3, London
  - Research Site 1, Manchester
  - Research Site 4, Manchester
  - Research Site 2, Oxford
  - Research Site 6, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coombes RC, Howell S, Lord SR, Kenny L, Mansi J, Mitri Z, Palmieri C, Chap LI, Richards P, Gradishar W, Sardesai S, Melear J, O'Shaughnessy J, Ward P, Chalasani P, Arkenau T, Baird RD, Jeselsohn R, Ali S, Clack G, Bahl A, McIntosh S, Krebs MG. Dose escalation and expansion cohorts in patients with advanced breast cancer in a Phase I study of the CDK7-inhibitor samuraciclib. Nat Commun. 2023 Jul 24;14(1):4444. doi: 10.1038/s41467-023-40061-y. PMID 37488191
- [Derived] Sava GP, Fan H, Coombes RC, Buluwela L, Ali S. CDK7 inhibitors as anticancer drugs. Cancer Metastasis Rev. 2020 Sep;39(3):805-823. doi: 10.1007/s10555-020-09885-8. PMID 32385714